CLINICAL TRIAL: NCT03245762
Title: Intranasal Oxytocin for Treatment of Infants and Children With Prader-Willi Syndrome in Nutritional Phase 1a - Phase 2 Study
Brief Title: Intranasal Oxytocin for Infants With Prader-Willi Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Prader-Willi Syndrome Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB201700423 -A; OCR16237 (Other: University of Florida)
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Results first posted 2019-06-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: This will be a double-blinded study, as no studies to date have compared this treatment in infants with placebo. Board-certified speech and language pathologist who will be blinded to the treatment arm of each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal oxytocin (Active Comparator): Intervention: 4 IU/day of intranasal oxytocin via a nasal spray device each morning.
  Interventions: Drug: Oxytocin
- IN-placebo (Placebo Comparator): Intervention: 4 IU/day of placebo via nasal spray device each morning.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 4 IU/day of oxytocin administered via nasal spray device each morning.
  Other Names: Syntocinon
  Arms: Intranasal oxytocin
Drug: Placebo — 4 IU/day of placebo administered via nasal spray device each morning
  Other Names: Saline
  Arms: IN-placebo

SUMMARY:
The purpose of this study is to compare the change in suck and swallow competency from baseline to morning of day 6 with intranasal oxytocin spray vs placebo in infants/children with Prader-Willi Syndrome who are in nutritional phase 1a. Videofluoroscopic swallow studies will be performed on treatment day 1 and on the day following treatment morning of day 6.

DETAILED DESCRIPTION:
The overall objective of this Phase 2 trial is to compare the change from baseline to morning of day 6 of Internasal Oxytocin (IN-OT) on suck and swallow competency in infants/children with Prader-Willi Syndrome (PWS) who are in nutritional phase 1a.

Study Hypothesis 1: The Study team hypothesize that replacing Oxytocin (OT) in infants and children who are in nutritional phase 1a will improve their suck and swallow, potentially even eliminating the need for gastrostomy tubes and nasogastric tubes for feeding, and decreasing the risk of aspiration with oral feeding.

Study Hypothesis 2: The Study team hypothesize that replacing OT in infants and children with PWS will result in improved eye contact, daytime alertness, and feelings of bonding between the parents and the infant.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with genetically confirmed PWS who are in nutritional phase 1a, as determined by PI
2. Physical exam and laboratory results that are within the normal range.
3. Presence of a parent/caregiver/guardian that is able to consent for their participation.

Exclusion Criteria:

1. Exposure to any investigational agent in the 30 days prior to randomization.
2. Prior chronic treatment with oxytocin.
3. A medical condition that might interfere with the conduct of the study, confound interpretation of study results or endanger the subject's well-being.

Ages: 1 Week to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Miller, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intranasal Oxytocin | IN-placebo
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Oxytocin | IN-placebo | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 5 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 4 | 11
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 4 | 13
  Europe | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Suck and Swallow Competency in Infants/Children With PWS Who Are in Nutritional Phase 1a
Description: Swallow study Overall improvement
Time Frame: baseline to day 5
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Oxytocin | IN-placebo
Number analyzed (Participants) | 10 | 5
Participants
  Improved Competency | 8 | 4
  No Change in Competency' | 1 | 1
  Worsened Competency | 1 | 0
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs IN-placebo; Test type: Superiority; p = 0.930, Ordinal Categorical Analysis; Odds Ratio (OR) = 0.9

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Intranasal Oxytocin | IN-placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

LIMITATIONS AND CAVEATS:
Short study with small number of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT03245762/Prot_SAP_000.pdf